CLINICAL TRIAL: NCT00416481
Title: Development of a Geriatric Assessment Measure for Older Patients With Cancer
Brief Title: Assessing Older Patients With Cancer
Status: Completed | Type: Observational
Sponsor: Alliance for Clinical Trials in Oncology (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: CALGB-360401; CALGB-360401; CDR0000523527 (Registry Identifier: NCI Physician Data Query)
Record Dates: First submitted 2006-12-27; First posted 2006-12-28 (Estimated); Last update posted 2016-07-13 (Estimated); Status verified 2016-07

CONDITIONS: Unspecified Adult Solid Tumor, Protocol Specific
Keywords: unspecified adult solid tumor, protocol specific

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patient assessment: Patients undergo assessments of cognition and performance status using the healthcare professional-rated Karnofsky performance scale. These assessments are performed by healthcare personnel. Body mass index and the percentage of unintentional weight loss and the number of falls in the past 6 months are also assessed.
  Patients also complete self-administered questionnaires that measure level of functioning and need for services. It also includes questionnaires that measure higher levels of physical functioning, performance related to survival and clinically significant illness and measures of comorbidity and the impact on daily activities. Lastly, questionnaires are administered to measure the impact of cancer on patients' social functioning and perceived availability of social support.
  Patients then begin planned treatment.
  Interventions: Behavioral: quality of life questionnaires

INTERVENTIONS:
Behavioral: quality of life questionnaires

SUMMARY:
RATIONALE: Questionnaires that measure the ability of older patients to think, learn, remember, and make judgments and carry out daily activities may improve the ability to plan treatment for patients with cancer.

PURPOSE: This clinical trial is studying ways to assess older patients with cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the feasibility of administration of the geriatric assessment in elderly patients with cancer.
* Determine the percentage of patients able to complete the self-administered portion of the geriatric assessment without assistance.
* Determine the length of time necessary to complete the geriatric assessment.
* Determine the variance and number of missing items.
* Assess patient satisfaction with the questionnaire by identifying items that are distressing or difficult to comprehend.
* Assess the percentage of geriatric assessments that contain all three of the following items: Timed Up and Go Assessment, Blessed Orientation-Memory-Concentration Test, and healthcare professional-rated Karnofsky performance status.

Secondary

* Determine the proportion of patients who are able to complete the self-report portion of the questionnaire without assistance and the length of time needed to complete the geriatric assessment within patients of various sociodemographic factors and educational status.

OUTLINE: This is a multicenter study. Patients are stratified according to age (65 to 69 years vs 70 years and over).

Patients undergo assessments of cognition using the Blessed Orientation-Memory-Concentration Test; functional status using the Timed Up and Go Assessment (measures physical mobility); and performance status using the healthcare professional-rated Karnofsky performance scale. These assessments are performed by healthcare personnel. Body mass index and the percentage of unintentional weight loss and the number of falls in the past 6 months are also assessed.

Patients also complete the following self-administered questionnaires: Instrumental Activities of Daily Living (measures level of functioning and need for services); Activities of Daily Living (measures higher levels of physical functioning); Karnofsky Self-Reported Performance Rating Scale (related to survival and clinically significant illness); Physical Health Section of the Older American Resources and Services Questionnaire (measures comorbidity and the impact on daily activities); Hospital Anxiety and Depression Scale; Medical Outcomes Study (MOS) Social Activity Limitations Measure (measures the impact of cancer on patients' social functioning); and MOS Social Support Survey Emotional/Information and Tangible Subscales (measures perceived availability of social support).

Patients then begin planned treatment.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed malignancy at any stage
* Enrolled on any cooperative group-sponsored cancer treatment trial (treatment has not yet started), including trials on the Cancer Trials Support Unit

PATIENT CHARACTERISTICS:

* Any performance status allowed
* Must be able to follow directions in English
* Sufficient cognitive and psychological function to give consent

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Patients aged 65 years and older with a histologically confirmed malignancy enrolled on any cooperative group-sponsored cancer treatment trial.
Sampling Method: Non-Probability Sample
Enrollment: 93 (Actual)
Dates: Start 2006-12; Primary Completion 2011-10 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
Mean and median time to complete the entire geriatric assessment | Up to 3 years
Mean number of missing items in each subscale and the distribution of missing items | Up to 3 years
Percentage of patients who identify a scale to be upsetting or difficult to understand | Up to 3 years
Percentage of Geriatric Assessments for which all three items (Timed Up and Go Assessment, Blessed Orientation-Memory-Concentration Test, and the healthcare professional-rated Karnofsky performance status) are completed | Up to 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Alice B. Kornblith, PhD, Study Chair — Dana-Farber Cancer Institute
Locations (13):
- United States (13):
  - Elkhart General Hospital, Elkhart, Indiana
  - Howard Community Hospital, Kokomo, Indiana
  - Center for Cancer Therapy at LaPorte Hospital and Health Services, La Porte, Indiana
  - CCOP - Northern Indiana CR Consortium, South Bend, Indiana
  - Memorial Hospital of South Bend, South Bend, Indiana
  - Michiana Hematology-Oncology, PC - South Bend, South Bend, Indiana
  - Saint Joseph Regional Medical Center, South Bend, Indiana
  - Lakeland Regional Cancer Care Center - St. Joseph, Saint Joseph, Michigan
  - University Medical Center of Southern Nevada, Las Vegas, Nevada
  - CCOP - Nevada Cancer Research Foundation, Las Vegas, Nevada
  - CCOP - Hematology-Oncology Associates of Central New York, East Syracuse, New York
  - Duke Comprehensive Cancer Center, Durham, North Carolina
  - Arthur G. James Cancer Hospital and Richard J. Solove Research Institute at Ohio State University Comprehensive Cancer Center, Columbus, Ohio

REFERENCES:
- [Result] Hurria A, Cirrincione CT, Muss HB, Kornblith AB, Barry W, Artz AS, Schmieder L, Ansari R, Tew WP, Weckstein D, Kirshner J, Togawa K, Hansen K, Katheria V, Stone R, Galinsky I, Postiglione J, Cohen HJ. Implementing a geriatric assessment in cooperative group clinical cancer trials: CALGB 360401. J Clin Oncol. 2011 Apr 1;29(10):1290-6. doi: 10.1200/JCO.2010.30.6985. Epub 2011 Feb 28. PMID 21357782